CLINICAL TRIAL: NCT07386093
Title: The Effect of Skin Color Scale Material Used by Families at Home in the Postnatal Period on the Process of Hospital Admission Due to Jaundice and Breastfeeding Parameters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Neva Çöpden, midwife, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: IUC-GEI-NC-01
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Neonatal Jaundice
Keywords: newborn; neonatal jaundice
MeSH Terms: conditions — Jaundice, Neonatal | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The Skin Color Scale Material (S-CARD / Neonatal Jaundice Monitoring Card) developed by the researcher and its user guide will be provided; verbal and visual training on the use of the material will be provided. Parents will be asked to observe their baby's skin color for the first 7 days after birth and record it on the monitoring card.
Who Masked: Care Provider
Masking Description: Families in this group will only receive routine, verbal information from the unit upon discharge. Both groups will be monitored similarly, but training on the use of the Skin Color Scale Material (S-CARD / Neonatal Jaundice Monitoring Card) will only be given to the experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The group using the Skin Color Scale Material (S-CARD / Neonatal Jaundice Monitoring Card). (Experimental): The Skin Color Scale Material (S-CARD / Neonatal Jaundice Monitoring Card) developed by the researcher and its user guide will be provided; verbal and visual training on the use of the material will be provided. Parents will be asked to observe their baby's skin color for the first 7 days after birth and record it on the monitoring card.
  Interventions: Other: Experiment Group
- Group not using Skin Color Scale Material (S-CARD / Neonatal Jaundice Monitoring Card) (Active Comparator): Families in this group will only receive routine, verbal information from the unit upon discharge. Both groups will be monitored similarly, but training on the use of the Skin Color Scale Material (S-CARD / Neonatal Jaundice Monitoring Card) will only be given to the experimental group.
  Interventions: Other: control group

INTERVENTIONS:
Other: Experiment Group — The Skin Color Scale Material (S-CARD / Neonatal Jaundice Monitoring Card) developed by the researcher and its user guide will be provided; verbal and visual training on the use of the material will be provided. Parents will be asked to observe their baby's skin color for the first 7 days after birth and record it on the monitoring card.
  Arms: The group using the Skin Color Scale Material (S-CARD / Neonatal Jaundice Monitoring Card).
Other: control group — Families in this group will only receive routine, verbal information from the unit upon discharge. Both groups will be monitored similarly, but training on the use of the Skin Color Scale Material (S-CARD / Neonatal Jaundice Monitoring Card) will only be given to the experimental group.
  Arms: Group not using Skin Color Scale Material (S-CARD / Neonatal Jaundice Monitoring Card)

SUMMARY:
The aim of this research is to evaluate the effect of the Skin Color Scale Material used by families in the postnatal period on the hospital admission process due to jaundice and breastfeeding parameters.

Although neonatal jaundice is mostly physiological, it can lead to serious complications such as kernicterus if not detected in time. Visually supported educational materials developed to provide early awareness can help families both to regularly monitor the baby's skin color and to notice the signs of jaundice in time.

DETAILED DESCRIPTION:
The Skin Color Scale Material (S-CARD / Neonatal Jaundice Monitoring Card), developed within the scope of this study, is a unique material based on visual assessment of skin color. The material includes 6 color ranges adapted from the Bili-ruler reference, with spaces reserved for observation and guiding statements to indicate the risk level opposite each color. With these features, it makes it possible for parents and healthcare professionals to easily visually detect jaundice. A user guide has also been prepared to support the correct and safe use of the card. The guide, which includes 6 instructions explaining the use of the card step by step and 5 warning notes for possible symptoms, not only provides a visual scale but also functions as a user-friendly and reliable guide. The research will be conducted through experimental and control groups determined by random assignment. Parents in the experimental group will be given detailed information about the use of the Skin Color Scale Material (S-CARD / Neonatal Jaundice Monitoring Card); Parents will be asked to observe their babies' skin color daily for the first 7 days after birth and compare their observations with the card. The control group will only receive standard verbal information at discharge, as already applied in the unit. In both groups, breastfeeding parameters (frequency, duration, general condition after breastfeeding) will be monitored on the 3rd and 7th days after discharge. The sample of the study consists of newborns with a birth weight ≥2500 grams, born between 36-42 weeks, without multiple pregnancies, and at least one parent who is literate, along with their parents. Participant selection will be made from among newborns and parents who meet the eligibility criteria. Data will be collected using the Personal Information Form, Newborn Monitoring Form, Skin Color Scale Material (S-CARD / Newborn Jaundice Monitoring Card), Parent Opinion Assessment Form, and Bristol Breastfeeding Assessment Tool developed by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born alive between 36-42 weeks of gestation or delivered healthy to their mothers,
* Newborns with a birth weight of 2500 grams or more,
* Newborns without a history of multiple pregnancy (twins, triplets, etc.),
* Newborns with at least one literate parent,
* Newborns whose families voluntarily agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Newborns younger than 36 weeks and requiring intensive care, or newborns older than 42 weeks,
* Newborns weighing less than 2500 grams at birth,
* Newborns requiring postnatal intensive care,
* Newborns with congenital anomalies, metabolic diseases, or serious clinical problems,
* Newborns whose families wish to withdraw from the study during the follow-up period or whose contact information is unavailable,
* Newborns excluded from analysis due to incomplete or erroneous data,
* Newborns whose families did not sign the informed consent form.

Ages: 36 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Data Collection Form | One month
  Developed by the researcher and their consultant in line with the literature (source). It is a form consisting of 34 questions. Participants' demographic characteristics, obstetric history, and information regarding childbirth will be obtained through this form.

SECONDARY OUTCOMES:
Bristol Lactation Assessment Tool (BEDS) | one month
  This is a form developed by Jenny Ingram in 2014 and validated in Turkish by Dolgun et al. in 2018. The application time for the scale is 5-10 minutes. While the Cronbach alpha value of the original form of the instrument was found to be 0.68, it was found to be 0.77 in the Turkish adaptation study. Scoring of the scale:
  Each item is scored between 0-2 points. The lowest score obtained from the scale is 0, and the highest score is 8. It will be used to evaluate the breastfeeding success of babies. This instrument covers parameters such as breastfeeding frequency, duration, time of initiation of breastfeeding, and the general condition of the baby.
Newborn Monitoring Form | one month
  This is a chart consisting of 7 questions developed by the researcher and their advisor in line with the literature. Data regarding the clinical follow-up period of the infants included in the study will be recorded in this form.
S-card Parent Feedback Evaluation Form: | one month
  It is a form consisting of 14 questions developed by the researcher and his/her advisor in line with the literature.

IPD SHARING:
Plan to Share IPD: No